CLINICAL TRIAL: NCT06112158
Title: The Effect of Web-Assisted Peer Education for Early Diagnosis of Breast Cancer on Health Beliefs, Knowledge Levels and Breast Self-Examination in University Students
Acronym: Early Diagnosi
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Esra ÖZER (Other)
Collaborators: Ankara Medipol University (Other)
Responsible Party: Sponsor-Investigator, Esra ÖZER, Assist. Proff., Ankara Medipol University
Organization: Ankara Medipol University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Screening
Other Study IDs: AMU-SBF-EO-131
Record Dates: First submitted 2023-10-27; First posted 2023-11-01 (Actual); Last update posted 2024-03-15 (Actual); Status verified 2024-03

CONDITIONS: University Students; Breast Self-examination; Health Education
Keywords: Breast self-examination; Health Education; University students; Breast cancer
MeSH Terms: conditions — Breast Self-Examination; Health Education; Breast Neoplasms | interventions — Early Intervention, Educational

STUDY DESIGN:
Intervention Model Description: Two groups with randomized controlled trial
Who Masked: Participant
Masking Description: Web-supported and face-to-face training on breast cancer information and screening will be provided to the experimental group.and outcome assessments will be performed by a investigator who was blinded to group allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education Intervention (Experimental): The BSE training program for the early diagnosis of breast cancer will be offered to students in two ways: face-to-face and via web support.
  While the training program prepared by the researchers was applied to the intervention group, it was planned that no application would be applied to the nonınterventıon group.
  In this study, the training period was determined in two ways:
  First; In face-to-face training, each training is planned as four sessions of 45 minutes. Each session is planned with a different purpose and application.
  Latter; The system will continue to be open during the training provided through web support and face-to-face training, but the system will be closed to access immediately after the face-to-face training is completed.
  Interventions: Behavioral: Education Intervention
- nonıntervention Group (No Intervention): Until the research is finalized, no intervention will be made. After the research is finalized, the system will be opened to the nonınterventıon group and the university in general to contribute to their knowledge and awareness.

INTERVENTIONS:
Behavioral: Education Intervention — The BSE training program for the early diagnosis of breast cancer will be offered to students in two ways: face-to-face and via web support.
  Content of training Session 1: Topics such as the structure of the breast, the definition of breast cancer, its prevalence, risk factors and symptoms Session 2: Teaching the importance of early diagnosis in breast cancer, the importance and benefits of BSE, the technique of performing BSE, the obstacles to the application of BSE.
  Session 3: Teaching the risk factors that cause breast cancer. Session 4: Discussion of case reports of patients diagnosed with breast cancer. Supporting education with web support
  Arms: Education Intervention

SUMMARY:
The aim of this study was to examine the effect of web-supported peer education on health beliefs, knowledge levels and breast self-examination in university students.

DETAILED DESCRIPTION:
In line with the general purpose of the study, an experimental design will be used in the study. The population of this study consists of female students of Ankara Medipol University. Considering that there may be dropouts from the study in line with the determined sample size, 200 students (intervention; n=100, control; n=100) who were excluded from the exclusion criteria and who agreed to participate in the study were planned to constitute the study group.

Hypotheses of the Research Between the experimental group and the control group, which received peer education on breast cancer and Breast Self-Examination (BSE); H1a1: There is a difference in terms of the sensitivity subscale score average. H1b1: There is a difference in terms of the mean score of the seriousness/importance subscale.

H1c1: There is a difference in terms of the average score of the benefit perception subscale.

H1d1: There is a difference in terms of the average score of the obstacle perception subscale.

H1e1: There is a difference in terms of the mean score of the trust subscale. H1f1: There is a difference in terms of the health motivation subscale score average.

H2a1: There is a difference in terms of the average knowledge score. H3a1: There is a difference in terms of performing breast self-examination.

ELIGIBILITY:
Inclusion Criteria:

* Young women who do not have any diagnosis of cancer or breast cancer
* who have no communication barriers
* who are not pregnant or breastfeeding
* who volunteer to participate in the study

Exclusion Criteria:

* Participants with a previous cancer diagnosis
* CHCMM training and who were absent for more than two sessions in the intervention group

Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2024-03-13 (Actual); Primary Completion 2024-05-30 (Estimated); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Comprehensive Breast Cancer Information Test | four months
  Questions from 1 to 12 on the scale; general knowledge about breast cancer; Questions 13 to 20 contain information about the treatability of breast cancer. It also consists of 20 questions that can be answered as "true" or "false". 1 point for each correct answer given; 0 points are given for incorrect answers and blank items. As the score obtained from the scale increases, the level of knowledge also increases.
Champion Health Belief Model Scale | four months
  It is used to determine women's beliefs and attitudes about breast cancer and breast self-examination. Each sub-dimension of the scale is evaluated separately. Champion Health Belief Model Scale (CHBMS) has 6 subscales and is a 5-point Likert type. "Perception of sensitivity" (3 items), "perception of seriousness" (7 items), "perception of benefit" (4 items), "perception of obstacle" (11 items), "trust" (10 items), "Health" regarding breast cancer It has sub-dimensions "motivation" (7 items). The total score of the scale is not calculated. Receiving a low score on the "obstacle perception" subscale and a high score on other subscales shows that women have positive attitudes and beliefs about breast cancer and breast self-examination practices.
Breast self-examination proficiency rating instrument-BSEPRI | four months
  This form was used to assess women's ability to perform breast self-examination according to the appropriate stages and their ability to find breast masses. In the form, there are 10 statements including the stages of performing CHBM. Each stage of the examination that is performed correctly is given 10 points, and 0 points are given for incorrect or non-performed stages. Accordingly, a minimum of 0 and a maximum of 100 points are obtained from the form. A score of 90 and above indicates that "CHCMM is performed correctly" and a score of 80 and below indicates that "CHCMM is not performed correctly".

SECONDARY OUTCOMES:
Semi-structured Interview Form | four months
  "Can you tell us about how the training has changed your life?", "What has this training added to your knowledge about breast cancer and CHCMM?", "What are the beneficial aspects of this training?" and "What are the aspects of this training that need to be improved?".

CONTACTS AND LOCATIONS:
Locations (1):
- Ankara Medipol Unıversty, Ankara, Turkey (Türkiye)